CLINICAL TRIAL: NCT03198845
Title: Therapeutic Effects Video Game Play Therapy on Patients With Knee Osteoarthritis: a Single Blind, Randomized-controlled Clinical Trial
Brief Title: Effects of Video Game on Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST 103-2314-B-341-002
Record Dates: First submitted 2017-06-23; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis; video game; therapeutic effects
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video game (Active Comparator): Participants received a total of twelve 40-min sessions of hot pack therapy combined transcutaneous electrical nerve simulation over the knees followed by 20-min supervised video game play therapy 20-min per session for 3 times per week for a 4-week duration.
  Therapeutic effects of video game intervention for patients with knee osteoarthritis were assessed.
  Interventions: Other: video game
- exercise group (Sham Comparator): Participants received a total of twelve 40-min sessions of hot pack therapy combined transcutaneous electrical nerve simulation over the knees followed by 20-min supervised therapeutic exercise 20-min per session for 3 times per week for a 4-week duration.
  Therapeutic effects of therapeutic exercise for patients with knee osteoarthritis were assessed.
  Interventions: Other: exercise

INTERVENTIONS:
Other: video game — 20-min per session for 3 times per week for a 4-week duration
  Arms: video game
Other: exercise — 20-min per session for 3 times per week for a 4-week duration
  Arms: exercise group

SUMMARY:
To investigate the effects of video game play therapy in patients with knee osteoarthritis

DETAILED DESCRIPTION:
A total of 80 patients with knee osteoarthritis were randomized into two groups, including video game group and exercise group.

Physical activity, quality of life, emotion, and balance were assessed at before treatment and follow-up assessments, including at after 2 week of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis with Kellgren/Lawrence grade II of greater ambulatory for more than 15 meters without support or orthosis usage

Exclusion Criteria:

* Knee operation history participants with pregnancy stroke history infection or fracture over lower limbs previously

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
change of Western Ontario and McMaster Universities Osteoarthritis index | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Western Ontario and McMaster Universities Osteoarthritis index

SECONDARY OUTCOMES:
change of quality of life | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  World Health Organization-Quality of life-Brief Vision
change of emotion | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Hospital Anxiety and Depression Scale
change of fatigue | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Multidimensional Fatigue Inventory

OTHER OUTCOMES:
change of disability | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Graded chronic pain scale
change of work ability | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Work ability index
change of balance | scores change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  Biodex Stability System
change of stairs climbing time | time change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  stairs climbing time
change of walking time | time change from baseline to after 2 weeks of treatment; after 4 weeks of treatment; and 1 and 3 months after treatment is terminated.
  walking 10-m time

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No